CLINICAL TRIAL: NCT06223919
Title: Randomized Trial to Evaluate the Efficacy/Effectiveness, Safety, and Immunogenicity of Replicative Live Attenuated Vaccinia Virus Vaccine LC16m8 for Prevention Against Mpox in High-risk Populations During Vaccination Deployment in Colombia
Brief Title: Efficacy/Effectiveness, Safety, and Immunogenicity of LC16m8 Mpox Vaccine in Colombia
Acronym: MPOX-COL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Collaborators: Ministerio de Salud y Protección Social de Colombia (Unknown); Ministry of Health, Labour and Welfare, Japan (Other Government); Japan Agency for Medical Research and Development (Other Government); National Center for Global Health and Medicine, Japan (Other Government); National Institute of Infectious Disease, Japan (Unknown); Instituto Nacional de Salud (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI-UN-1760
Record Dates: First submitted 2023-12-28; First posted 2024-01-25 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Monkeypox
Keywords: Vaccines; monkeypox; Mpox; Mpox virus
MeSH Terms: conditions — Mpox, Monkeypox | interventions — smallpox vaccine LC16m8

STUDY DESIGN:
Intervention Model Description: Vaccinate LC16m8 randomly assigned to two groups consisting of two groups of Immediate and Delayed vaccination 1:1 with a follow-up period of 180 days to evaluate newly MPXV-infected cases as well as immuno-responses including neutralizing antibody titers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate vaccination (Experimental): This vaccin is a yellowish-yellow dry preparation containing live vaccinia virus (strain LC16m8). When the accompanying solvent is added, it dissolves rapidly to form a clear or slightly cloudy yellowish-red or reddish liquid. The ingredients of this vaccin are contained in 0.5 mL of a solution of this product dissolved in 0.5 mL of the accompanying solvent (20 vol% glycerin-added water for injection).
  Just one dose of vaccine will be administered according to standardized operating procedure (SOP). Briefly, the vaccine is dissolved with 0.5 mL of a diluent provided. The reconstituted vaccine is usually administered percutaneously at a dose of approximately 0.025 mL by the multiple puncture technique using a bifurcated needle. The number of punctures will be 15 times. Procedures for vaccine administration are described in detail in the SOP. The participant must be observed at the vaccination site for 30 minutes after vaccine administration to observe possible immediate reactions.
  Interventions: Biological: LC16m8
- Delayed vaccination (Active Comparator): The use of placebo as a control group is essential to scientifically assess the efficacy of vaccines in clinical trials and to obtain reliable evidence in preventing the onset of disease. However, the use of a placebo is unethical. Subjects are at high risk of mpox and must not be given a placebo. Therefore, a design was applied in which the immediate treatment group was evaluated with the delayed group as a control group. A period of six weeks was set aside between the immediate and delayed treatment groups to be used for logistics, such as preparations and delivery of the vaccine in the delayed treatment group. It is ethical, for the same reason, because it prevents inequities based on the abovementioned reasons.
  Interventions: Biological: LC16m8

INTERVENTIONS:
Biological: LC16m8 — LC16m8 should be stored at temperatures between -35°C and -20°C. The product should not be stored at temperatures below -35°C, because deterioration or damage of the rubber stopper could occur.
  The virus in this product is sensitive to sunlight and is quickly inactivated, so care should be taken to avoid exposure to light, both before or after reconstitution.
  Carefully examine the content at the time of reconstitution. Do not use if precipitation, contamination of foreign substances, or other abnormalities are observed.
  This product should be dissolving the drug immediately before inoculation. Once dissolved, it should be used immediately. Since this product does not contain thimerosal, once the stopper is removed, any solution remained in the vial must be disposed of.
  Do not restore or reuse the remaining solution. Shelf Life: 10 years from the date of passing the national test for lot-release Bottle containing about 250 doses

SUMMARY:
Background: Mpox is a zoonotic disease caused by the mpox virus (MPXV). It has been endemic in West and Central African countries. However, the soaring number of those has been reported in non-endemic countries since May 2022, making World Health Organization (WHO) declare a global mpox Public Health Emergency of International Concern in July 2022. Those with mpox are primarily young men (96%, and median age of 34 [interquartile range (IQR):29-41 years]), and 84% are self-identified homosexual, bisexual, and men who have sex with men (MSM) . Furthermore, about half of these mpox cases with known human immunodeficiency virus 1(HIV-1, hereafter shown as HIV). WHO recommended prioritizing vaccinating those populations as high-risk populations, including those with HIV, since they will be severely ill if infected mpox virus (MPXV). The smallpox vaccine is expected to offer cross-immunity against MPXV. Under these circumstances, WHO included LC16m8 in the recommended vaccine lists for mpox as the product is expected to have cross-efficacy and immunogenicity against MPXV. Additionally, the safety profile was demonstrated in both adults and children, including infants who have low immuno-functions. Given that Colombia has the fifth highest mpox prevalence worldwide, WHO encouraged the authorities to implement vaccine programs while evaluating the safety and efficacy of LC16m8 as collaborative research. Following WHO initiative, this study is being conducted with the collaboration of various experts from Colombia and Japan on a large scale, with vaccine contributions and funding from Japan and Colombia However, the current infection situation differs from six months ago, and there have been few recent cases of MPXV infection in the country.

Primary objective: To determine the efficacy of the replicating attenuated live vaccinia virus vaccine LC16m8 against laboratory-confirmed mpox and safety in a Colombian population with a high risk of being infected with MPXV(See the Inclusion Criteria), by comparing the immediate vaccination group and the delayed vaccination groups to assess safety and tolerability until 180 days after vaccination. Study design: An open randomized deployment study (1:1 Immediate and Delayed vaccination group).

Study population: People at high risk of serious illness if infected with MPXV and those who engage in risk behaviors for acquiring MPXV infection.

DETAILED DESCRIPTION:
Hypothesis: LC16m8 is a safe and effective vaccine for high-risk immunocompromised populations, including those living with HIV.

Intervention evaluation plan: Vaccinate with LC16m8 those people randomly assigned to two groups: immediate and deferred vaccination 1:1 with a follow-up period of 180 days to evaluate new cases infected by MPXV.

General design: This research is being carried out within the framework of the mpox vaccination implementation program in Colombia. It comprises the following three complementary components:

* Study section 1: Parallel open sequential randomized controlled trial to evaluate the efficacy of LC16m8 vaccine in preventing MPXV infection.
* Study section 2: Cohort study based on the same population base
* Study section 3: Cohort study compared to real world cohort

STUDY SECTION 1: Participants will receive LC16m8 vaccine within 6 weeks (immediate vaccination) or 6 weeks later (delayed vaccination) after randomization. Both groups will be followed up at 14, 30 and 180 days after vaccination, mainly through phone calls.

The study will compare the incidence of new MPXV infections in the early vaccination group from day 14 to day 42 after vaccination with the incidence of rate at which new MPXV infections occur in the delayed vaccination group from 42 days before to 14 days after vaccination; this comparison will be made from the hazard ratio or proportional hazard model.

Additionally, the immune response, including neutralizing antibody titers, will be evaluated from the day of vaccination (Day 1) to 180 days post-vaccination in 60 participants, who will be selected from a single research center and only belonging to the immediate vaccination group. Two 5 mL blood samples (converted to serum) will be collected from the participants for immunogenicity assessments at the following time points: Days 0, 14 (+/-2), 30 (+/-2), and 180 (+/-7) post-vaccination. Another blood sample for immunogenicity assessment will be collected before the vaccine is administered on Day 0.

Safety events will be intensively sought, especially in the first 14 days after vaccine administration and all those arising within 180 days post-vaccination. Participants will also self-report symptoms through a mobile application designed for this purpose.

STUDY SECTION 2 AND 3 (NESTED STUDIES)

- Study of cohorts supported on the same population base: A total of 1,000 vaccinated individuals, including participants in section 1 of the study, will make up the exposed group. The unexposed group will consist of 4,000 unvaccinated individuals from the same population base (a list of HIV patients with a CD4 count greater than 200 cells/ml and PrEP users). who are patients with HIV and CD4 greater than 200 cells/mm3, and PrEP users. The group of unvaccinated individuals are people who meet the study's criteria but did not agree to be vaccinated or withdrew their consent. We will compare the cumulative incidence of these two groups over a 180-day period. We will obtain information about non-participants and withdrawals from the records at the INS and local health entities. We will use the hazard ratio (HR) to compare these groups, and we will also conduct a propensity score analysis.The objective is to demonstrate the effectiveness and safety of the LC16m8 replicating vaccine against laboratory-confirmed MPXV in a Colombian population at high risk of MPXV infection (see inclusion criteria).

Assumptions:

* A relative risk reduction (RRR) of 75% is assumed to calculate the sample size.
* Confidence level: 95%
* Ratio of vaccinated:unvaccinated: 1:4

  * RRR: Risk (Rx) in the unvaccinated group - Rx in the vaccinated group/(Rx) in the unvaccinated group.

The incidence of the event (Mpox case) is considered to be 0.4% per period in the exposed group (I Exp (+)) and 1.6% per period in the unexposed group (I exp (-)), in accordance with the current situation of Mpox infection in Colombia.

Incidence in vaccinated 4/1000 = 0.004 Incidence in unvaccinated 64/4000 = 0.016 RR** = 0.2756 (95% CI: 0.1057 ; 0.7185) **Relative risk (RR): Risk (Rx) in unvaccinated/Rx in vaccinated RAR***: -1.2888 (95% CI: -2.247; - 0.3306) RRR= 0.7244 (95% CI: 0.2815; 0.8943) Power: 0.92 where RR is relative risk, RAR is absolute risk reduction and RRR is relative risk reduction.

The Ho could be rejected.

- Cohort study compared to the real-world cohort: There will be no sample size because all the information from the databases will be used in the cohort, so a sample is not necessary since we will take all the subjects in HIV and PrEP programs.

ELIGIBILITY:
1. Inclusion Criteria:

   1. Sex: Males and females
   2. Age: ≥18 and ≤ 50 years old
   3. Persons must be willing and sign the Informed Consent (I.C.).
   4. Any of the following conditions including clinical conditions /manifestation:

      * People living with the HIV, with stable infection determined by participant´s being on antiretroviral therapy with a blood CD4+ cell count, ≥ 200 cells/mm3 in the last six months before study enrolment
   5. Persons that use PrEP (HIV Pre-exposure prophylaxis).
   6. Homosexual, Bisexual, or other men who have sex with men (MSM) with multiple sexual partners. Commercial sex workers (CSW) and partners CSW
   7. A female participant is eligible to participate if the participant meets one of the inclusion criteria numbered -1, -2 or -3 above. The participant cannot be pregnant or lactating. Additionally, the female participant must meet one of the following conditions:

      * The participant has non-childbearing potential. To be considered of non-childbearing potential, a female must be post-menopausal for at least one year or surgically sterile. OR
      * The participant has a childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks before the vaccine administration until at least 2 months after the administration and have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) within 10 days before vaccination.
2. Exclusion Criteria:

   1. Subjects with an unstable medical condition as determined by their initial medical history, physical examination, or laboratory results
   2. Subjects with a terminal disease.
   3. Subjects with a medical record of anaphylaxis caused by any of the vaccine's excipients or with previous undesired reactions to other vaccines such us (Allergic reactions, Guillain barre syndrome, Varicella zoster, or shingles).
   4. Previous medical record of Mpox.
   5. Subjects living with HIV with a CD4+ T cell count of fewer than 200 cells/mm3.
   6. Pregnant or breastfeeding woman.
   7. Active or medical record of atopic dermatitis or eczema, or with close contact with someone with an active or medical record of atopic dermatitis or eczema.
   8. The presence of a skin condition with extensive breaks in the skin, such as burns, impetigo, contact dermatitis, or zoster (shingles), is not likely to heal by the day of vaccination.
   9. Using immunosuppressive medications, in eye drops, by mouth, or topically (nasal sprays and inhaled corticosteroids are permissible).
   10. Active or past malignancy except for cutaneous basal or squamous cell carcinomas.
   11. An Autoimmune disease.
   12. History of heart failure with decreased left ventricular ejection fraction (<40%).
   13. Medical record of splenectomy.
   14. Medical record of solid organ or bone marrow transplantation.
   15. Medical record of keloid scar development
   16. Psychiatric condition that precludes compliance with the protocol.
   17. People who received or plan to receive licensed live vaccines 30 days before or after study vaccination.
   18. People who received or planned to receive immunoglobulin or other blood products 60 days before HIV screening.
   19. People who received or plan to receive experimental drugs/vaccines 30 days before study vaccination or before study completion.
   20. People who received or planned to receive systemic immunosuppressive therapy and radiation therapy 30 days before or after the study vaccination.
   21. Use of systemic chemotherapy within five years before the study vaccination.
   22. Medical record of smallpox vaccination and/or evidence of scarring at the vaccination site.
   23. Allergies to streptomycin sulfate and/or erythromycin lactobionate.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8686 (Estimated)
Dates: Start 2023-12-16 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of mpox infection between the immediate versus delayed vaccination groups from day 15 to day 56 post-vaccination of the immediate group. | For immediate vaccination group: from days 15th to 56th post vaccination. For delayed vaccination group: from enrollment to the day of vaccination (42 days later)
  The incidence rate of new cases of mpox (laboratory-confirmed) will be calculated with a 95% confidence interval (CI) based on the Poisson distribution for each vaccination group. The time to the onset of the first occurrence of a confirmed mpox case in the subject will be summarized graphically using the Kaplan-Meier method.
Incidence of adverse events between the vaccination groups | up to 6 months post vaccination
  Proportion of adverse events (serious and non-serious) presented in participants included in the two vaccination groups (immediate and delayed)
Incidence rate of mpox infection between the vaccinated cohort versus the unvaccinated cohort | 6 months post vaccination
  The incidence rate of new cases of mpox (laboratory-confirmed) will be calculated with a 95% confidence interval (CI) based on the Poisson distribution for each cohort. The time to the onset of the first occurrence of a confirmed mpox case in the subject will be summarized graphically using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Frequency of laboratory-confirmed severe cases of MPOX in the immediate and delayed vaccination groups. | 6 months post-vaccination
  Proportion of participants with confirmed MPOX that presented severe symptoms requiring hospitalization, emergency department care, or death associated with MPOX.
Incidence rate of mpox suspected cases without laboratory confirmation between the immediate versus delayed vaccination groups from day 15 to day 56 post-vaccination of the immediate group. | - For immediate vaccination group: from days 15th to 56th post vaccination. For delayed vaccination group: from enrollment to the day of vaccination (42 days later
  Mpox suspected cases correspond to participants that present with skin lesions to the emergency room or treating patient.
Proportion of patients with seroconversion of geometric mean neutralizing titer (GMT) of LC16m8. | up to 6 months post vaccination
  Seroconversion is considered in cases where the titer on day 30 is 4 times higher than on day 0.
Geometric mean of LC16m8 neutralizing titer by vaccination group. | up to 6 months post vaccination
  overall geometric mean of each group (immediate and delayed vaccination)
Geometric mean of LC16m8 neutralizing titer by helper T lymphocytes (CD4) count in each vaccination group | up to 6 months post vaccination
  Subgroups of patients with a CD4 count of 350 or less and those with a CD4 count greater than 350 will be compared for each vaccination group.
Maximum lesion area (MLA) in mm² after scarification with vaccination LC16m8 | up to 6 months post vaccination
  take area measured 14 days post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Álvarez, Principal Investigator — Universidad Nacional de Colombia
Locations (3):
- Colombia (3):
  - Clinica Universitaria Colombia - Centro Medico Teusaquillo, Bogotá, Bogota D.C.
  - Hospital Universitario San Ignacio, Bogotá, Bogota D.C.
  - Infecto Clinicos, Bogotá, Bogota D.C.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adnan N, Haq ZU, Malik A, Mehmood A, Ishaq U, Faraz M, Malik J, Mehmoodi A. Human monkeypox virus: An updated review. Medicine (Baltimore). 2022 Sep 2;101(35):e30406. doi: 10.1097/MD.0000000000030406. PMID 36107544
- [Background] Karagoz A, Tombuloglu H, Alsaeed M, Tombuloglu G, AlRubaish AA, Mahmoud A, Smajlovic S, Cordic S, Rabaan AA, Alsuhaimi E. Monkeypox (mpox) virus: Classification, origin, transmission, genome organization, antiviral drugs, and molecular diagnosis. J Infect Public Health. 2023 Apr;16(4):531-541. doi: 10.1016/j.jiph.2023.02.003. Epub 2023 Feb 9. PMID 36801633
- [Background] Mitja O, Ogoina D, Titanji BK, Galvan C, Muyembe JJ, Marks M, Orkin CM. Monkeypox. Lancet. 2023 Jan 7;401(10370):60-74. doi: 10.1016/S0140-6736(22)02075-X. Epub 2022 Nov 17. PMID 36403582
- [Background] Di Giulio DB, Eckburg PB. Human monkeypox: an emerging zoonosis. Lancet Infect Dis. 2004 Jan;4(1):15-25. doi: 10.1016/s1473-3099(03)00856-9. PMID 14720564
- [Background] Shchelkunov SN, Marennikova SS, Moyer RW. Orthopoxviruses pathogenic for humans: Springer Science & Business Media; 2006.
- [Background] McInnes et al. Family: Poxviridae [Website]. International Committee on Taxonomy of Viruses (ICTV); 2023 [updated 2023/04/17.
- [Background] Parker S, Buller RM. A review of experimental and natural infections of animals with monkeypox virus between 1958 and 2012. Future Virol. 2013 Feb 1;8(2):129-157. doi: 10.2217/fvl.12.130. PMID 23626656
- [Background] Magnus Pv, Andersen EK, Petersen KB, Birch-Andersen A. A POX-LIKE DISEASE IN CYNOMOLGUS MONKEYS. Acta Pathologica Microbiologica Scandinavica. 1959;46(2):156-76.
- [Background] Kozlov M. Monkeypox in Africa: the science the world ignored. Nature. 2022 Jul;607(7917):17-18. doi: 10.1038/d41586-022-01686-z. No abstract available. PMID 35739391
- [Background] Tomori O, Blumberg L. Response to the multi-country monkeypox outbreak: a view from Africa. J Travel Med. 2022 Dec 27;29(8):taac138. doi: 10.1093/jtm/taac138. No abstract available. PMID 36440640
- [Background] Esposito JJ, Knight JC. Orthopoxvirus DNA: a comparison of restriction profiles and maps. Virology. 1985 May;143(1):230-51. doi: 10.1016/0042-6822(85)90111-4. PMID 2998003
- [Background] Likos AM, Sammons SA, Olson VA, Frace AM, Li Y, Olsen-Rasmussen M, Davidson W, Galloway R, Khristova ML, Reynolds MG, Zhao H, Carroll DS, Curns A, Formenty P, Esposito JJ, Regnery RL, Damon IK. A tale of two clades: monkeypox viruses. J Gen Virol. 2005 Oct;86(Pt 10):2661-2672. doi: 10.1099/vir.0.81215-0. PMID 16186219
- [Background] Bunge EM, Hoet B, Chen L, Lienert F, Weidenthaler H, Baer LR, Steffen R. The changing epidemiology of human monkeypox-A potential threat? A systematic review. PLoS Negl Trop Dis. 2022 Feb 11;16(2):e0010141. doi: 10.1371/journal.pntd.0010141. eCollection 2022 Feb. PMID 35148313
- [Background] Velavan TP, Meyer CG. Monkeypox 2022 outbreak: An update. Trop Med Int Health. 2022 Jul;27(7):604-605. doi: 10.1111/tmi.13785. Epub 2022 Jun 14. No abstract available. PMID 35633308
- [Background] Edouard Mathieu FS, Saloni Dattani, Hannah Ritchie and Max Roser -
- [Background] WHO. Multi-country outbreak of mpox, External situation report #19 - 30 March 2023 2023 [Available from: https://www.who.int/publications/m/item/multi-country-outbreak-of-mpox--external-situation-report--19---30-march-2023.
- [Background] Mitja O, Alemany A, Marks M, Lezama Mora JI, Rodriguez-Aldama JC, Torres Silva MS, Corral Herrera EA, Crabtree-Ramirez B, Blanco JL, Girometti N, Mazzotta V, Hazra A, Silva M, Montenegro-Idrogo JJ, Gebo K, Ghosn J, Pena Vazquez MF, Matos Prado E, Unigwe U, Villar-Garcia J, Wald-Dickler N, Zucker J, Paredes R, Calmy A, Waters L, Galvan-Casas C, Walmsley S, Orkin CM; SHARE-NET writing group. Mpox in people with advanced HIV infection: a global case series. Lancet. 2023 Mar 18;401(10380):939-949. doi: 10.1016/S0140-6736(23)00273-8. Epub 2023 Feb 21. PMID 36828001
- [Background] Farahat RA, Abdelaal A, Shah J, Ghozy S, Sah R, Bonilla-Aldana DK, Rodriguez-Morales AJ, McHugh TD, Leblebicioglu H. Monkeypox outbreaks during COVID-19 pandemic: are we looking at an independent phenomenon or an overlapping pandemic? Ann Clin Microbiol Antimicrob. 2022 Jun 15;21(1):26. doi: 10.1186/s12941-022-00518-2. No abstract available. PMID 35706004
- [Background] Nalca A, Rimoin AW, Bavari S, Whitehouse CA. Reemergence of monkeypox: prevalence, diagnostics, and countermeasures. Clin Infect Dis. 2005 Dec 15;41(12):1765-71. doi: 10.1086/498155. Epub 2005 Nov 11. PMID 16288402
- [Background] Yon H, Shin H, Shin JI, Shin JU, Shin YH, Lee J, Rhee SY, Koyanagi A, Jacob L, Smith L, Lee SW, Rahmati M, Ahmad S, Cho W, Yon DK. Clinical manifestations of human Mpox infection: A systematic review and meta-analysis. Rev Med Virol. 2023 Jul;33(4):e2446. doi: 10.1002/rmv.2446. Epub 2023 Apr 13. PMID 37056203
- [Background] WHO. Multi-country monkeypox outbreak: situation update; 27 June 2022 2022 [Available from: https://www.who.int/emergencies/disease-outbreak-news/item/2022-DON396.
- [Background] Poland GA, Kennedy RB, Tosh PK. Prevention of monkeypox with vaccines: a rapid review. Lancet Infect Dis. 2022 Dec;22(12):e349-e358. doi: 10.1016/S1473-3099(22)00574-6. Epub 2022 Sep 15. PMID 36116460
- [Background] WHO. Laboratory testing for the monkeypox virus. Interim guidance 23 May 2022 2022 [Available from: https://www.who.int/publications-detail-redirect/WHO-MPX-laboratory-2022.1.
- [Background] Fine PE, Jezek Z, Grab B, Dixon H. The transmission potential of monkeypox virus in human populations. Int J Epidemiol. 1988 Sep;17(3):643-50. doi: 10.1093/ije/17.3.643. PMID 2850277
- [Background] Siegrist EA, Sassine J. Antivirals With Activity Against Mpox: A Clinically Oriented Review. Clin Infect Dis. 2023 Jan 6;76(1):155-164. doi: 10.1093/cid/ciac622. PMID 35904001
- [Background] WHO. Background document for the SAGE October 2022 session on monkeypox vaccines 2022 [Available from: https://www.who.int/publications/i/item/WHO-MPX-Immunization.
- [Background] KM Biologics Co. L. Maximizing the Use of Freeze-Dried Smallpox Vaccine Prepared in Cell Culture LC16 "KMB" in Emergencies. 2023.
- [Background] SOCIAL MDSYP. VIRUELA SIMICA; MONKEYPOX 2023 [Available from: https://app.powerbi.com/view?r=eyJrIjoiNjQzZGQ0ZjAtODRhMi00MzFhLWFmODctOWMxNGVkNGFjMDhkIiwidCI6ImE2MmQ2YzdiLTlmNTktNDQ2OS05MzU5LTM1MzcxNDc1OTRiYiIsImMiOjR9
- [Background] WHO. Multi-country outbreak of mpox; External Situation Report, published 11 May 2023 2023 [Available from: https://www.who.int/publications/m/item/multi-country-outbreak-of-mpox--external-situation-report--22---11-may-2023.
- [Background] UNAIDS. AIDS HIV Estimate; Colombia [Available from: https://www.unaids.org/en/regionscountries/countries/colombia.
- [Background] Cuenta de Alto Costo (CAC) FCdEdAC, Cuenta de Alto Costo (CAC). . Situación del VIH en Colombia 2022; Bogotá, D.C. 2023) [Available from: https://cuentadealtocosto.org/site/vih/vih-sida-en-colombia-retos-y-apuestas-en-salud/.
- [Background] Johnson PLF, Bergstrom CT, Regoes RR, Longini IM, Halloran ME, Antia R. Evolutionary consequences of delaying intervention for monkeypox. Lancet. 2022 Oct 8;400(10359):1191-1193. doi: 10.1016/S0140-6736(22)01789-5. Epub 2022 Sep 21. No abstract available. PMID 36152668
- [Background] Morales-Zamora G, Espinosa O, Puertas E, Fernandez JC, Hernandez J, Zakzuk V, Cepeda M, Alvis-Guzman N, Castaneda-Orjuela C, Paternina-Caicedo A. Cost-Effectiveness Analysis of Strategies of COVID-19 Vaccination in Colombia: Comparison of High-Risk Prioritization and No Prioritization Strategies With the Absence of a Vaccination Plan. Value Health Reg Issues. 2022 Sep;31:101-110. doi: 10.1016/j.vhri.2022.04.004. Epub 2022 May 26. PMID 35640462
- [Background] Kenner J, Cameron F, Empig C, Jobes DV, Gurwith M. LC16m8: an attenuated smallpox vaccine. Vaccine. 2006 Nov 17;24(47-48):7009-22. doi: 10.1016/j.vaccine.2006.03.087. Epub 2006 Apr 21. PMID 17052815
- [Background] Hirayama M. In search of attenuated vaccine. Clinical special edition: vaccination in future-everything about attenuated vaccine. Rinsho to Uirusu [Clin Virus]. 1975;3:225-8.
- [Background] Hashizume S. Properties of attenuated mutant of vaccinia virus, LC16m8, derived from Lister strain. Vaccinia Viruses as Vectors for Vaccine Antigens. 1985:87-99.
- [Background] Hashizume S. Basics of New Attenuated Vaccine Strain LC16m8. Clinic and Virus ,1975 1975;Vol 3 No . 33:,229・35.
- [Background] Saijo M, Ami Y, Suzaki Y, Nagata N, Iwata N, Hasegawa H, Ogata M, Fukushi S, Mizutani T, Sata T, Kurata T, Kurane I, Morikawa S. LC16m8, a highly attenuated vaccinia virus vaccine lacking expression of the membrane protein B5R, protects monkeys from monkeypox. J Virol. 2006 Jun;80(11):5179-88. doi: 10.1128/JVI.02642-05. PMID 16698998
- [Background] Iizuka I, Ami Y, Suzaki Y, Nagata N, Fukushi S, Ogata M, Morikawa S, Hasegawa H, Mizuguchi M, Kurane I, Saijo M. A Single Vaccination of Nonhuman Primates with Highly Attenuated Smallpox Vaccine, LC16m8, Provides Long-term Protection against Monkeypox. Jpn J Infect Dis. 2017 Jul 24;70(4):408-415. doi: 10.7883/yoken.JJID.2016.417. Epub 2016 Dec 22. PMID 28003603
- [Background] Gordon SN, Cecchinato V, Andresen V, Heraud JM, Hryniewicz A, Parks RW, Venzon D, Chung HK, Karpova T, McNally J, Silvera P, Reimann KA, Matsui H, Kanehara T, Shinmura Y, Yokote H, Franchini G. Smallpox vaccine safety is dependent on T cells and not B cells. J Infect Dis. 2011 Apr 15;203(8):1043-53. doi: 10.1093/infdis/jiq162. PMID 21450994
- [Background] Yokote H, Shinmura Y, Kanehara T, Maruno S, Kuranaga M, Matsui H, Hashizume S. Safety of attenuated smallpox vaccine LC16m8 in immunodeficient mice. Clin Vaccine Immunol. 2014 Sep;21(9):1261-6. doi: 10.1128/CVI.00199-14. Epub 2014 Jul 2. PMID 24990910
- [Background] Yokote H, Shinmura Y, Kanehara T, Maruno S, Kuranaga M, Matsui H, Hashizume S. Vaccinia virus strain LC16m8 defective in the B5R gene keeps strong protection comparable to its parental strain Lister in immunodeficient mice. Vaccine. 2015 Nov 9;33(45):6112-9. doi: 10.1016/j.vaccine.2015.07.076. Epub 2015 Aug 1. PMID 26241947
- [Background] Yamaguchi M, Kimura M, Hirayama M. Vaccination research group research report: Ministry of Health and Welfare special research: postvaccination side effects and research regarding treatment of complications. Rinsho To Uirusu. 1975;3:269-79.
- [Background] Kennedy JS, Gurwith M, Dekker CL, Frey SE, Edwards KM, Kenner J, Lock M, Empig C, Morikawa S, Saijo M, Yokote H, Karem K, Damon I, Perlroth M, Greenberg RN. Safety and immunogenicity of LC16m8, an attenuated smallpox vaccine in vaccinia-naive adults. J Infect Dis. 2011 Nov;204(9):1395-402. doi: 10.1093/infdis/jir527. Epub 2011 Sep 15. PMID 21921208
- [Background] Pharmaceutical Safety and Environmental Health Bureau、Pharmaceutical Evaluation Division. Report on the Deliberation Results. 2022.
- [Background] Nishiyama Y, Fujii T, Kanatani Y, Shinmura Y, Yokote H, Hashizume S. Freeze-dried live attenuated smallpox vaccine prepared in cell culture "LC16-KAKETSUKEN": Post-marketing surveillance study on safety and efficacy compliant with Good Clinical Practice. Vaccine. 2015 Nov 9;33(45):6120-7. doi: 10.1016/j.vaccine.2015.09.067. Epub 2015 Oct 9. PMID 26455406
- [Background] Saito T, Fujii T, Kanatani Y, Saijo M, Morikawa S, Yokote H, Takeuchi T, Kuwabara N. Clinical and immunological response to attenuated tissue-cultured smallpox vaccine LC16m8. JAMA. 2009 Mar 11;301(10):1025-33. doi: 10.1001/jama.2009.289. PMID 19278946
- [Background] Sanz-Munoz I, Sanchez-dePrada L, Sanchez-Martinez J, Rojo-Rello S, Dominguez-Gil M, Hernan-Garcia C, Fernandez-Espinilla V, de Lejarazu-Leonardo RO, Castrodeza-Sanz J, Eiros JM. Possible Mpox Protection from Smallpox Vaccine-Generated Antibodies among Older Adults. Emerg Infect Dis. 2023 Mar;29(3):656-658. doi: 10.3201/eid2903.221231. Epub 2023 Feb 2. PMID 36732061
- [Background] Crum-Cianflone NF, Wallace MR. Vaccination in HIV-infected adults. AIDS Patient Care STDS. 2014 Aug;28(8):397-410. doi: 10.1089/apc.2014.0121. Epub 2014 Jul 16. PMID 25029589
- [Background] Overton ET, Stapleton J, Frank I, Hassler S, Goepfert PA, Barker D, Wagner E, von Krempelhuber A, Virgin G, Meyer TP, Muller J, Badeker N, Grunert R, Young P, Rosch S, Maclennan J, Arndtz-Wiedemann N, Chaplin P. Safety and Immunogenicity of Modified Vaccinia Ankara-Bavarian Nordic Smallpox Vaccine in Vaccinia-Naive and Experienced Human Immunodeficiency Virus-Infected Individuals: An Open-Label, Controlled Clinical Phase II Trial. Open Forum Infect Dis. 2015 May 5;2(2):ofv040. doi: 10.1093/ofid/ofv040. eCollection 2015 Apr. PMID 26380340
- [Background] FDA. FACT SHEET FOR HEALTHCARE PROVIDERS ADMINISTERING VACCINE: EMERGENCY USE AUTHORIZATION OF JYNNEOS (SMALLPOX AND MONKEYPOX VACCINE, LIVE, NON-REPLICATING) FOR PREVENTION OF MONKEYPOX DISEASE IN INDIVIDUALS DETERMINED TO BE AT HIGH RISK FOR MONKEYPOX INFECTION 2022 [Available from: https://www.fda.gov/media/160774/download.
- [Background] Geretti AM, Brook G, Cameron C, Chadwick D, French N, Heyderman R, Ho A, Hunter M, Ladhani S, Lawton M, MacMahon E, McSorley J, Pozniak A, Rodger A. British HIV Association Guidelines on the Use of Vaccines in HIV-Positive Adults 2015. HIV Med. 2016 Aug;17 Suppl 3:s2-s81. doi: 10.1111/hiv.12424. No abstract available. PMID 27568789
- [Background] Banaszkiewicz A, Radzikowski A. Efficacy, effectiveness, immunogenicity--are not the same in vaccinology. World J Gastroenterol. 2013 Nov 7;19(41):7217-8. doi: 10.3748/wjg.v19.i41.7217. PMID 24222970
- [Background] Curran KG, Eberly K, Russell OO, Snyder RE, Phillips EK, Tang EC, Peters PJ, Sanchez MA, Hsu L, Cohen SE, Sey EK, Yin S, Foo C, Still W, Mangla A, Saafir-Callaway B, Barrineau-Vejjajiva L, Meza C, Burkhardt E, Smith ME, Murphy PA, Kelly NK, Spencer H, Tabidze I, Pacilli M, Swain CA, Bogucki K, DelBarba C, Rajulu DT, Dailey A, Ricaldi J, Mena LA, Daskalakis D, Bachmann LH, Brooks JT, Oster AM; Monkeypox, HIV, and STI Team. HIV and Sexually Transmitted Infections Among Persons with Monkeypox - Eight U.S. Jurisdictions, May 17-July 22, 2022. MMWR Morb Mortal Wkly Rep. 2022 Sep 9;71(36):1141-1147. doi: 10.15585/mmwr.mm7136a1. PMID 36074735
- [Background] WHO. Vaccines and immunization for monkeypox: Interim guidance, 16 November 2022 2022 [Available from: https://www.who.int/publications/i/item/WHO-MPX-Immunization.
- [Background] VIH PCd. Prep-Colombia.org [Available from: https://prep-colombia.org/como-funciona/.
- [Background] WHO. Strategic Preparedness, Readiness and Response Plan, MONKEYPOX 2022 [Available from: https://www.who.int/publications/m/item/monkeypox-strategic-preparedness--readiness--and-response-plan-(sprp).
- [Background] Social MdSyP. Guía de Práctica Clínica (GPC) basado en la evidencia científica para la atención de la infeccion por VIH/SIDA en personas adultas, gestantes y adolescentes (Clinical Practice Guideline based on scientific evidence for the care of HIV/AIDS infection in adults, pregnant women and adolescents) 2021 [Available from: https://www.minsalud.gov.co/sites/rid/Lists/BibliotecaDigital/RIDE/INEC/IETS/gpc-vih-adultos-2021.pdf.
- [Background] Mbala PK, Huggins JW, Riu-Rovira T, Ahuka SM, Mulembakani P, Rimoin AW, Martin JW, Muyembe JT. Maternal and Fetal Outcomes Among Pregnant Women With Human Monkeypox Infection in the Democratic Republic of Congo. J Infect Dis. 2017 Oct 17;216(7):824-828. doi: 10.1093/infdis/jix260. PMID 29029147
- [Background] Reed JL, Scott DE, Bray M. Eczema vaccinatum. Clin Infect Dis. 2012 Mar;54(6):832-40. doi: 10.1093/cid/cir952. Epub 2012 Jan 30. PMID 22291103
- [Background] KMB. Package Insert: Freeze-dried Smallpox Vaccine Prepared in Cell Culture LC16m8 (KMB). 2022.
- [Background] World Health Organization. WHO declares the end of the monkeypox emergency and calls for sustained efforts for the long-term management of the disease [Internet]. World Health Organization; May 2023 Available at: https://www.paho.org/es/noticias/11-5-2023-oms-declara-fin-emergency-por-viruela-simica-pide-esfuerzos-sostenidos-para
- [Background] Henao-Restrepo AM, Camacho A, Longini IM, Watson CH, Edmunds WJ, Egger M, Carroll MW, Dean NE, Diatta I, Doumbia M, Draguez B, Duraffour S, Enwere G, Grais R, Gunther S, Gsell PS, Hossmann S, Watle SV, Konde MK, Keita S, Kone S, Kuisma E, Levine MM, Mandal S, Mauget T, Norheim G, Riveros X, Soumah A, Trelle S, Vicari AS, Rottingen JA, Kieny MP. Efficacy and effectiveness of an rVSV-vectored vaccine in preventing Ebola virus disease: final results from the Guinea ring vaccination, open-label, cluster-randomised trial (Ebola Ca Suffit!). Lancet. 2017 Feb 4;389(10068):505-518. doi: 10.1016/S0140-6736(16)32621-6. Epub 2016 Dec 23. PMID 28017403
- [Background] Hoffmann C, Jessen H, Wyen C, Grunwald S, Noe S, Teichmann J, Krauss AS, Kolarikal H, Scholten S, Schuler C, Bickel M, Roll C, Kreckel P, Koppe S, Straub M, Klausen G, Lenz J, Esser S, Jensen B, Rausch M, Unger S, Pauli R, Harter G, Muller M, Masuhr A, Schafer G, Seybold U, Schellberg S, Schneider J, Monin MB, Wolf E, Spinner CD, Boesecke C. Clinical characteristics of monkeypox virus infections among men with and without HIV: A large outbreak cohort in Germany. HIV Med. 2023 Apr;24(4):389-397. doi: 10.1111/hiv.13378. Epub 2022 Sep 4. PMID 36059149
- [Background] EMA. Classification and analysis of the GCP inspection findings of GCP inspections conducted at the request of the CHM (Inspection reports to EMA 2000-2012) 2014 [updated 01 December 204. Available at: https://www.ema.europa.eu/en /documents/other/classification-analysis-good-clinical-practice-gcp-inspection-findings-gcp-inspections-conducted_en.pdf.
- [Background] Austin PC. Balance diagnostics for comparing the distribution of baseline covariates between treatment groups in propensity-score matched samples. Stat Med. 2009 Nov 10;28(25):3083-107. doi: 10.1002/sim.3697. PMID 19757444
- [Background] Austin PC, Small DS. The use of bootstrapping when using propensity-score matching without replacement: a simulation study. Stat Med. 2014 Oct 30;33(24):4306-19. doi: 10.1002/sim.6276. Epub 2014 Aug 4. PMID 25087884